CLINICAL TRIAL: NCT05320497
Title: Application of Transparent Cap-assisted Digital Cholangioscopy (SpyGlassTM) for Biliary Stricture
Brief Title: Transparent Cap-assisted SpyGlass for Biliary Stricture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Transparent Cap
Record Dates: First submitted 2022-03-21; First posted 2022-04-11 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Bile Duct Stricture; Endoscopic Retrograde Cholangiopancreatography; Biliary Disease; Biliary Tract Neoplasms
Keywords: Bile Duct Stricture; ERCP; Choledochoscopy; Transparent Cap; Biliary biopsy
MeSH Terms: conditions — Gallbladder Diseases; Biliary Tract Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a before-after study. Transparent cap SpyGlass and standard SpyGlass were performed on the same patient successively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transparent cap-assisted SpyGlass (Experimental): Add a transparent cap to the end of the SpyGlass choledochoscopy
  Interventions: Device: Transparent cap

INTERVENTIONS:
Device: Transparent cap — Add a self-made transparent cap (made by cutting a silicone drainage tube) to the end of the SpyGlass choledochoscope, and then perform routine choledochoscopy and biopsy operations

SUMMARY:
The transparent cap-assisted endoscope has the function of fixing field of view and increasing visual space. It has been widely used in gastrointestinal examination and treatment. In this study, the investigators intend to apply transparent cap-assisted choledochoscopy to endoscopic biliary tract exploration and biopsy to investigate whether transparent cap-assisted choledochoscopy can improve operability, visual field clarity, and biopsy accuracy.

DETAILED DESCRIPTION:
Recently, endoscopy has become more widely used in clinical practice. A straightforward method of improving mucosal visualization involves attachment of a transparent cap to the end of the endoscope. It has been widely used in gastrointestinal examination and treatment.This is a before-after study. In patients with suspected bile duct stricture, tandem ERCP combined with SpyGlass choledochoscopy procedures were carried out on the same day in random order, first without a transparent cap and then with a cap (without-to-with), or first with a cap and then without a cap (with-to-without). The differences in maneuverability, visual field clarity and biopsy accuracy of choledochoscopy with and without transparent cap were recorded to explore the application prospect of transparent cap assisted choledochoscopy.

ELIGIBILITY:
Inclusion Criteria:

* The indications for ERCP.
* Written informed consent

Exclusion Criteria:

* Underlying bleeding disorder
* The platelet count less than 50×10^9/L
* Serious cardio-pulmonary, hepatic or renal disease
* Intolerance to ERCP
* Other high-risk conditions or disease (such as massive ascites, etc.)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-07-10 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The clearness of visual field | Immediately
  The clearness of visual field was evaluated by the operating physician and was rated as "clear" or "not clear."
Intubation rates of bile duct ends, cystic duct openings, and left and right hepatic duct bifurcations | Immediately
  Comparison of intubation rates between transparent cap SpyGlass and standard SpyGlass

SECONDARY OUTCOMES:
Biopsy accuracy | 1 week
  Biopsy accuracy between clear cap SpyGlass and standard SpyGlass was evaluated by comparing the coincidence rate of biopsy histopathology and postoperative pathology

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of Chinese PLA General Hosptial, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No